CLINICAL TRIAL: NCT00035087
Title: An Open-Label Phase IIa Trial Evaluating the Safety and Efficacy of EPO906 as Therapy in Patients With Advanced Colorectal Cancer
Brief Title: EPO906 Therapy in Patients With Advanced Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEPO906A2201
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Colorectal Neoplasms; Colonic Neoplasms
Keywords: colon; rectum; colorectal; rectal; cancer; tumor; tumour; neoplasm; carcinoma; intravenous; epothilone
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Neoplasms; Carcinoma | interventions — epothilone B

INTERVENTIONS:
Drug: epothilone b

SUMMARY:
This study will examine whether the new investigational drug EPO906, given by intravenous infusion (IV directly into the vein), is effective in shrinking tumors and preventing the growth of cells that cause colorectal cancer.

ELIGIBILITY:
Inclusion Criteria

Patients must meet the following criteria to be eligible for the study:

* Histologically or cytologically documented evidence of colorectal cancer with at least one measurable lesion (if previous radiation treatment, the target lesion must have demonstrated progression since the radiation)
* The patient should have failed or progressed on no more than two prior chemotherapies for metastatic disease (the prior chemotherapy must have included a fluoropyrimidine and either Irinotecan or oxaliplatin, or any combination of these agents, with the last chemotherapy having contained Irinotecan or oxaliplatin)
* Patients who have received only adjuvant therapy for their disease are eligible, as long as they have relapsed within six months of completing such therapy and that therapy contained 5-FU and Irinotecan or oxaliplatin administered in combination as part of an investigational protocol
* Must have a life expectancy of greater than three (3) months.

Exclusion Criteria

The following patients are not eligible for the study:

* Patients with symptomatic CNS metastases or leptomeningeal involvement
* Patients with unresolved bowel obstruction
* Patients with any peripheral neuropathy or unresolved diarrhea greater than Grade 1
* Patients with severe cardiac insufficiency
* Patients who have undergone major surgery for any cause less than 4 weeks prior to study entry
* Patients with radiation therapy or chemotherapy within the last four weeks
* Patients taking Coumadin or other warfarin-containing agents with the exception of low dose Coumadin (1 mg or less) for the maintenance of in-dwelling lines or ports
* History of another malignancy within 5 years prior to study entry except curatively treated non-melanoma skin cancer or cervical cancer in situ
* Patients with active or suspected acute or chronic uncontrolled infection including abcesses or fistulae
* HIV+ patients
* Pregnant or lactating females

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2002-05; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Tumor response as assessed by radiologic techniques and/or physical examination based on Response Evaluation Criteria in Solid Tumors (RECIST)

SECONDARY OUTCOMES:
Time to progression
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Cancer Institute of New Jersey (CINJ), New Brunswick, New Jersey, United States